CLINICAL TRIAL: NCT03828942
Title: Monitoring the HeMAtological TOXicity of Drugs
Brief Title: Monitoring the HeMAtological TOXicity of Drugs (HeMATOX)
Acronym: HeMATOX
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Joe Elie Salem, Assistant director, clinical investigation center Paris Est, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-19-01
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Hematological Abnormality; Hematotoxicity
Keywords: advrese event; hematotoxicity; drugs; chemotherapies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Hematological toxicity induced by drugs and chemotherapies: Case reported in the World Health Organization (WHO) of hematological toxicities of patient treated by a drug, with a chronology compatible with the drug toxicity
  Interventions: Drug: drug inducing hematological toxicity

INTERVENTIONS:
Drug: drug inducing hematological toxicity — Drugs susceptible to induce hematological toxicities

SUMMARY:
Several drugs and chemotherapies seem to have an impact on the hematological system. This study investigates reports of hematological toxicities, including the International classification of disease ICD-10 for treatments in the World Health Organization (WHO) global Individual Case Safety Report (ICSR) database (VigiBase).

DETAILED DESCRIPTION:
Several drugs and chemotherapies seem to have an impact on the hematological system and are responsible of a wide range of hematological side effects. Those are poorly described, due to the modification of the pharmacopeia, and the recent recognition of several of these adverse events. This study investigates the main characteristics of patients affected by rare hematological side effects imputed to drugs. A causality assessment according to the WHO-UMC (World Health Organization - Uppsala Monitoring Center) is systematically applied.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the WHO's pharmacovigilance database till 01/02/2019

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with a drug that could be reported in the WHO's pharmacovigilance database
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2023-04-08 (Actual)

PRIMARY OUTCOMES:
Hematological toxicities of drugs Identification and report of cases of hematological toxicities associated with drugs. | to 01/02/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports

SECONDARY OUTCOMES:
Causality assessment of reported hematological toxicities events according to the WHO system | to 01/02/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
Description of the type of hematological toxicity depending on the category of drug | to 01/02/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
Description of the other immune related adverse events concomitant to the hematological toxicity induced by drugs | to 01/02/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
Description of the duration of treatment when the toxicity happens (role of cumulative dose) | to 01/02/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
Description of the drug-drug interactions associated with adverse events | to 01/02/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
Description of the pathologies (cancer) for which the incriminated drugs have been prescribed | to 01/02/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
Description of the population of patients having hematological toxicity adverse event | to 01/02/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM, Paris
  - Rhumatology department, CHU Strasbourg, Hautepierre hospital, Strasbourg

IPD SHARING:
Plan to Share IPD: Undecided